CLINICAL TRIAL: NCT01735903
Title: Objective Measures of Nerve Integrity, Posture, Gait and Blood Flow, After Nerve Decompression In diabetiC Neuropathy PatiENTs
Brief Title: Objective Measures of Nerve Integrity, Posture, Gait and Blood Flow, After Nerve Decompression
Acronym: OMNIFICENT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Foot Surgery Center of Northern Colorado (Other)
Collaborators: Association of Extremity Nerve Surgeons (Other)
Responsible Party: Principal Investigator, James Anderson, DPM, Principal Investigator, Foot Surgery Center of Northern Colorado
Other Study IDs: OMNI1
Record Dates: First submitted 2012-11-15; First posted 2012-11-28 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Diabetic Peripheral Neuropathy
MeSH Terms: interventions — Gait

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Arm A - Non-Diabetic, Gait and Balance — Arm A will enroll patients WITHOUT diabetes, but with peripheral neuropathy and lower limb pain, paresthesia, gait disturbances, or motor weakness and will follow the same protocol except the subject will NOT participate in blood flow testing performed at Colorado State University, and therefore do not include the inclusion/exclusion criterion that are specifically related to the blood flow assessment.
  Subjects may have any combination of lower limb nerve decompression surgery of the listed surgical sites with or without the addition of Soleal Sling Decompression. Soleal Sling Decompression surgical procedure will require the use of a thigh tourniquet.

SUMMARY:
The purpose of this study is to measure the effect of nerve decompression on the recovery of the treated nerves. To obtain objective data during surgery of the treated nerves' via electrical signals and muscle power when stimulated. Also, to monitor muscle strength, balance/gait and blood flow in the lower extremity before and after surgery.

DETAILED DESCRIPTION:
Nerve decompression (ND)as treatment for the foot complications of diabetic sensorimotor peripheral neuropathy (DSPN) is a controversial topic although many patients find it provides gratifying relief of pain and numbness. Neural electrical monitoring has been used intra-operatively to diagnosis nerve abnormality, monitoring for ongoing normal nerve function and confirm nerve integrity for spine surgeries and thyroid surgeries with success. Presently there is not objective data to indicate the the use of neural electrical monitoring is reliable or effective. The goal of this study is to measure objectively and quantifiable clinical surgical outcomes of nerve decompression surgery in diabetic neuropathy patients. The study is designed to measure changes in nerve function, gait, balance and blood flow in the lower limb.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with diabetic peripheral neuropathy and has nerve deficit in all proposed surgical areas, sensory and/or motor
* Patient has a positive provocative (i.e. Tinel's sign) observed clinically in the popliteal and tibial nerve trees.
* Patient is between 18 years and 85 years of age
* Patient is a type I or type II diabetic that is currently under medical treatment
* Patient has a Hgb A1C lab value of 8.0% or less
* Patient symptom based VAS scale is 6 or above for at least one of the following: pain, burning, numbness, tingling, weakness or instability
* Patient is scheduled for surgery and has been cleared for outpatient surgery per anesthesia guidelines established for the Foot Surgery Center of Northern Colorado
* Patient is able and willing to comply with all study requirements, including the follow-up evaluations and will return to the investigational site for all required office visits and CSU visits
* Patient has been informed of the nature of the study, agrees to its provisions and has provided written consent

Exclusions Criteria:

* Patient has a BMI of greater than 40 or body weight greater than 300 pounds
* Patient has untreated hypertension (systolic blood pressure > 160 and/or diastolic > 100)
* Patient's ASA is 4 or greater
* Patient has blood glucose greater than 200 the day of surgery
* Patient has Raynaud's Syndrome
* Patient is a current smoker
* Patient is a woman who is considering pregnancy or who is pregnant
* Patient has history of recent nerve or lumbar disc surgery, untreated thyroid disease, B12 or Folate deficiency, hepatic disease, renal disease, and/or Parkinson's disease, or neuropathy due to chemotherapy or radiation therapy
* Patient is being treated with chemotherapeutic agents
* Patient has ankle edema greater than mild - (Moderate to Severe)
* Patient is participating in another investigational device, biologic, or drug study and has not completed the primary endpoint(s) or if there is a potential for clinical interference beyond the primary endpoint

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Poudre Valley Foot and Ankle Clinic patients and Neuropathy Testing Center of Colorado
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-11; Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
EMG signals used intraoperative as objective measurements of change before and after nerve decompression surgery. Gait, balance and blood flow measurements before and after peripheral nerve decompression surgery | Within one month of surgical date, surgical date, 3 months and 6 months post operative or 4 months postoperative if the subjects elect to have the contralateral limb surgery prior to 3 months following the initial surgery.
  Primary Endpoint is assessed by changes in:
  * Neuromotor function in the lower limb as measured by intraoperative electromyographic(EMG) recordings of the muscles in the anterior and lateral compartments of the leg and muscles of the foot.
  * Blood flow in the lower limb both distal to and proximal to the nerve release sites, as measured by duplex doppler of the external femoral artery (a.), superficial femoral a., popliteal a., anterior and posterior tibial a., dorsal pedis a. Shear stress changes in these arteries.
  * Lower limb performance defined as:
  * Dorsiflexor strength and speed of contraction
  * Proprioception at the ankle
  * One-legged standing balance
  * Functional reach
  * Sensory function in the foot
  * Usual gait speed
  * Standardized tests of mobility

SECONDARY OUTCOMES:
Change in sensory perception | up to one month of surgical date, 3 months and 6 months post operative or 4 months postoperative if the subjects elect to have the contralateral limb surgery prior to 3 months following the initial surgery.
  * Two-point discrimination
  * Changes in nerve conduction measures
  * Changes in ankle-brachial index (ABI)
  * Visual Analog Score (VAS) for neuropathic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: James C. Anderson, DPM, Principal Investigator — Anderson Podiatry Center
Locations (1):
- Anderson Podiatry Center, Neuropathy Testing Center of Colorado, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided